CLINICAL TRIAL: NCT04846881
Title: A Phase III Randomized, Double-blind, Placebo-controlled, Parallel Group Trial to Examine the Efficacy and Safety of Iclepertin Once Daily Over 26 Week Treatment Period in Patients With Schizophrenia (CONNEX-2)
Brief Title: Clinical Trial of Iclepertin Effect on Cognition and Functional Capacity in Schizophrenia (CONNEX-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1346-0012; 2020-003744-84 (EudraCT Number)
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — BI 425809

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iclepertin 10 mg (Experimental): This arm comprised participants who received 10 mg tablet of iclepertin orally once daily, with doses administered at least 24 hours (hrs) apart, taken with water.
  Participants were treated for 26 weeks, followed by 4 weeks follow-up after trial drug termination.
  Interventions: Drug: Iclepertin
- Placebo (Placebo Comparator): This arm comprised participants who received 10 mg tablet of iclepertin-matched Placebo orally once daily, with doses administered at least 24 hrs apart, taken with water.
  Participants were treated for 26 weeks, followed by 4 weeks follow-up after trial drug termination.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iclepertin — One tablet of 10 mg iclepertin taken once daily for 26 weeks
  Other Names: BI 425809
  Arms: Iclepertin 10 mg
Drug: Placebo — One tablet of matching placebo taken once daily for 26 weeks
  Arms: Placebo

SUMMARY:
This study is open to adults with schizophrenia. Schizophrenia can affect the way a person thinks, their memory and their mental functioning. Examples include struggling to remember things, or to read a book or pay attention to a movie. Some people have difficulty calculating the right change or planning a trip so that they arrive on time. The purpose of this study is to find out whether a medicine called Iclepertin improves learning and memory in people with schizophrenia.

Participants are put into two groups randomly, which means by chance. One group takes Iclepertin tablets and the other group takes placebo tablets. Placebo tablets look like Iclepertin tablets but do not contain any medicine. Participants take a tablet once a day for 26 weeks. In addition, all participants take their normal medication for schizophrenia.

During this time, doctors regularly test learning and memory of the participants by use of questionnaires, interviews, and computer tests. The results of the mental ability tests are compared between the groups.

Participants are in the study for about 8 months. During this time, they visit the study site about 15 times and get about 3 phone calls from the study team. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria

1. Patient must be capable of providing a signed and dated written informed consent by visit 1 in accordance with International Council on Harmonisation for Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
2. Male or female patients who are 18-50 years (inclusive) of age at time of consent.
3. Diagnosis of schizophrenia utilizing Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) with the following clinical features:

   * Outpatient, clinically stable and in the residual (non-acute) phase of their illness.
   * No hospitalization3 or increase in level of psychiatric care4 due to worsening of schizophrenia within 12 weeks prior to randomization.
   * Positive and Negative Syndrome Scale (PANSS) score: items P1, P3-P6 = 5 and item P2 and P7 = 4 at Visit 1, and confirmed at Visit 2.
4. Patients should have functional impairment in day-to-day activities such as difficulties following conversation or expressing themselves, difficulties staying focused, difficulties remembering instructions, what to say or how to get to places, per investigator judgement.
5. Patients maintained on current antipsychotic treatment (minimum 1 and maximum 2 antipsychotics, but clozapine is not allowed) for at least 12 weeks and on current dose for at least 35 days prior to randomization.

   -- For patients on two antipsychotics, at least one antipsychotic must be within the approved label dose range. The second antipsychotic must not exceed the maximum daily dose per local label.

   Note: If the total dose is stable, different dosage forms of the same antipsychotic treatment will be considered as one antipsychotic.
6. Patients with any other concomitant psychoactive medications (except for anticholinergics) need to be maintained on same drug for at least 12 weeks and on current dose/ regimen for at least 35 days prior to randomization.

   * Maximum daily benzodiazepine load of up to 1 mg lorazepam-equivalent as needed.
   * For any other psychoactive medications cannot exceed the maximum daily dose per local label of the country where the study is being conducted.
7. Women of childbearing potential (WOCBP)5 must be ready and able to use highly effective methods of birth control per Non-Clinical Safety Studies for the Conduct of Human Clinical Trials and Marketing Authorization for Pharmaceuticals (ICH M3 (R2)) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the protocol. Such methods should be used throughout the trial, and for a period of at least 35 days after last trial drug intake, and the patient must agree to periodic pregnancy testing during participation in the trial.
8. Have a study partner, defined as any person either private or professional who knows the patient well, has been capable of interacting with the patient on regular basis, and preferably consistent throughout the study.

   * The study partner must interact with the patient at a minimum one hour per week and, preferably, at least 2 times a week. At least one interaction per week should be in person.
   * The study partner must have educational achievement of minimum 8th grade.
   * Professional study partners (e.g. study nurse, social worker etc.) are allowed if not involved in administration of any of the protocol assessments.

Further inclusion criteria apply.

Exclusion criteria

1. Patient with current DSM-5 diagnosis other than Schizophrenia, including but not limited to bipolar, schizoaffective, major depressive disorder etc. The Mini-International Neuropsychiatric Interview (M.I.N.I.) for psychotic disorders should be used for guidance.
2. Cognitive impairment due to developmental, neurological (e.g. stroke) or other disorders including head trauma, or patients with dementia or epilepsy.
3. Severe movement disorders

   * Leading to cognitive impairment (e.g. Parkinson's dementia), or
   * Interfering with the efficacy assessments, or
   * Due to antipsychotic treatment that cannot be controlled with low dose anticholinergic treatment (equal to maximum 1 mg benztropine twice daily).
4. Any suicidal behavior in the past 1-year prior to screening and during the screening period.
5. Suicidal ideation of type 5 in the Columbia Suicidality Severity Rating Scale (C-SSRS) (i.e. active suicidal thought with plan and intent) in the past 3 months prior to screening and up to and including Visit 2.

   -- Patients with Suicidal Ideation type 4 in the C-SSRS (i.e. active suicidal thought with intent but without specific plan), within 3 months prior to screening and up to and including visit 2, can be randomized in the study, if assessed and documented by a licensed mental health professional that there is no immediate risk of suicide.
6. History of moderate or severe substance use disorder (other than caffeine and nicotine), as defined in DSM-5 within the last 12 months prior to informed consent.
7. Positive urine drug screen at Visit 1 based on central lab test.
8. Patients who were treated with any of the following within 6 months prior to randomization:

   * Clozapine
   * Stimulants (e.g. methylphenidate, dextroamphetamine, modafinil)
   * Ketamine or esketamine
   * Electroconvulsive therapy (ECT) or modified ECT Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 611 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (127):
- United States (20):
  - Clinical Innovations, Inc, Bellflower, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - ASCLEPES Research Centers, P.C. dba Alliance Research, Long Beach, California
  - University of California Los Angeles, Los Angeles, California
  - NRC Research Institute, Orange, California
  - Collaborative Neuroscience Research, LLC-Torrance-69527, Torrance, California
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Research in Miami Inc, Hialeah, Florida
  - Optimus U Corporation-Miami-69452, Miami, Florida
  - Health Synergy Clinical Research, LLC, West Palm Beach, Florida
  - American Medical Research, Chicago, Illinois
  - Sheppard Pratt Physicians's Practice Association, Inc., Baltimore, Maryland
  - PsychCare Consultants Research, St Louis, Missouri
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - New York State Psychiatric Institute, New York, New York
  - Insight Clinical Trials, LLC, Independence, Independence, Ohio
  - Relaro Medical Trials, LLC, Dallas, Texas
  - John Peter Smith Health Network, Fort Worth, Texas
  - Salem VA Medical Center, Salem, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Argentina (8):
  - CENYDET-Centro Neurobiologico y de Estres Traumatico (Biopsychomedical Research Group S.R.L.), CABA
  - SERES Neurociencia Cognitiva Aplicada, CABA
  - Fundación FunDaMos para la asistencia e investigación en psiquiatría, CABA
  - CEN (Centro Especializado Neurociencias), Córdoba
  - Sanatorio Morra S.A., Córdoba
  - Clinica Privada de Salud Mental Santa Teresa de Avila, La Plata
  - Resolution Psychopharmacology Research Institute, Mendoza
  - Centro de Investigacion y Asistencia en Psiquiatria (CIAP), Rosario
- Brazil (5):
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Cpquali Pesquisa Clinica Ltda, São Paulo
  - Clínica Viver - Centro de Desospitalização Humana, São Paulo
  - Hospital das Clinicas da FMUSP, São Paulo
- Chile (2):
  - Biomedica Research Group, Santiago
  - Psicomed Estudios Clínicos, Segunda Región
- Croatia (5):
  - Clincal Hospital Centre Rijeka, Rijeka
  - Clinical Hospital Centre Zagreb, Zagreb
  - Solmed Polyclinic, Zagreb
  - Psychiatric Hospital 'Sveti Ivan', Zagreb
  - University Psychiatric Hospital Vrapce, Zagreb
- France (12):
  - HOP Charles Perrens, Bordeaux
  - HOP Gabriel-Montpied, Clermont-Ferrand
  - HOP Albert Chenevier, Créteil
  - HOP André Mignot, Le Chesnay-Rocquencourt
  - HOP Fontan, Lille
  - HOP la Colombière, Montpellier
  - HOP Hôtel-Dieu, Nantes
  - HOP Pasteur, Nice
  - HOP Carémeau, Nîmes
  - HOP Guillaume Régnier, Rennes
  - HOP Rouffach, Rouffach
  - HOP Nord-Saint-Priest-en-Jarez-53664, Saint-Priest-en-Jarez
- Hungary (4):
  - Obudai Egeszegugyi Centrum Kft., Budapest
  - Semmelweis University, Budapest
  - University of Debrecen, Gyula Kenezi University Hospital, Debrecen
  - PsychoTech Ltd., Pécs
- Japan (29):
  - Okehazama Hospital Fujita Kokoro Care Center, Aichi, Toyoake
  - Toyota Memorial Hospital, Aichi, Toyota
  - National Hospital Organization Shimofusa Psychiatric Medical Center, Chiba, Chiba
  - Uematsu Mental Clinic, Fukuoka, Chikugo
  - AK Clinic, Fukuoka, Fukuoka
  - Hirota Clinic, Fukuoka, Kurume
  - Kishi Hospital, Gumma, Kiryu
  - Hokudai-dori Mental Health Clinic, Hokkaido, Sapporo
  - Tatsuta Clinic, Hyogo, Kobe
  - Kanazawa Medical University Hospital, Ishikwa, Kahoku-gun
  - Kishiro Mental Clinic, Kanagawa, Kawasaki
  - Links Mental Clinic, Kanagawa, Yokohama
  - Yokohama City University Hospital, Kanagawa, Yokohama
  - Yuge Neuropsychiatric Hospital, Kumamoto, Kumamoto
  - Medical Corporation Yamadakai Yatsushiro Welfare Hospital, Kumamoto, Yatsushiro
  - Suwa Red Cross Hospital, Nagano, Suwa
  - Nara Medical University Hospital, Nara, Kashihara
  - University of the Ryukyus Hospital, Okinawa, Ginowan
  - Osaka City Hospital Organization Osaka City General Hospital, Osaka, Osaka
  - Rainbow and Sea Hospital, Saga, Karatsu
  - Inuo Hospital, Saga, Tosu
  - Medical Corporation Seijin Hospital, Tokyo, Adachi-ku
  - Institute of Science Tokyo Hospital, Tokyo, Bunkyo-ku
  - Nishigahara Hospital, Tokyo, Kita-ku
  - Minami-Aoyama Antique Street Clinic, Tokyo, Minato-ku
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - Maynds Tower Mental Clinic, Tokyo, Shibuya-ku
  - Shinjuku East Mental Clinic, Tokyo, Shinjuku-ku
  - Hokuriku Hospital, Toyama, Nanto
- Malaysia (4):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - University of Malaya Medical Centre, Kuala Lumpur
  - Hospital Sentosa, Kuching
  - Hospital Tuanku Ja'afar, Seremban, Negeri Sembilan
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastricht University, Maastricht
- Poland (7):
  - Psychiatric Doctor's Office Ireneusz Kaczorowski, Bełchatów
  - Podlassian Center of Psychogeriatry, Bialystok, Bialystok
  - Health Center Alcea, Gdansk
  - MentalMEDIC, Gliwice
  - Provincial Hospital for Nervous and Mentally Ill in Swiecie, Gmina Świecie
  - EUROMEDIS Sp. z o.o., Szczecin, Szczecin
  - Clinhouse, Zabrze
- Romania (2):
  - Mental Health Center Sector 4, Bucharest
  - SC Carpe Diem SRL, Sibiu
- Serbia (3):
  - Institute for Mental Health, Belgrade
  - Special Hospital for Psychiatric Diseases Sveti Vračevi, Novi Kneževac
  - Clinical Center of Vojvodina, Novi Sad
- Singapore (2):
  - Changi General Hospital, Singapore
  - Institute of Mental Health, Singapore
- Slovakia (3):
  - Psychiatria, Nemocnica s poliklinikou Prievidza so sidlom v Bojniciach, Bojnice
  - EPAMED s.r.o., Košice
  - Psychiatricka Ambulancia Psycholine s.r.o., Rimavská Sobota
- South Korea (5):
  - Inje University Haeundae Paik Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Hospital, Seoul
- Spain (13):
  - Hestia Palau, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario General de Villalba, Collado de Villalba
  - Hospital Universitario Reina Sofía, Córdoba
  - Centro de Salud mental de Getafe, Getafe
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital de Son Llàtzer, Palma
  - Centro de Salud de San Juan, Salamanca
  - Benito Menni Complejo Asistencial en Salud Mental, Sant Boi de Llobregat
  - Hospital Virgen del Rocío, Seville
  - Hospital Clinico Universitario De Valencia, Valencia
  - Hospital Nicolás Peña, Vigo
  - Hospital Provincial. Complejo Asistencial de Zamora, Zamora
- Communal Non-Profit Enterprise "Regional Clinical Psychiatric Hospital" of Kirovohrad Regional Council, Nove, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Keefe RSE, Harvey PD, Correll CU, Falkai P, Hashimoto N, Klein H, Krystal JH, Marder S, Medalia A, Sumiyoshi T, Wang G, Zhang H, Blahova Z, Bichard-Sall I, English BA, Fu E, Gruenenfelder F, Groeschl M, Kimura K, Tang W, von der Goltz C, Fowler C. Efficacy and safety of iclepertin for cognitive impairment associated with schizophrenia (CONNEX programme): results from three phase 3 randomised controlled trials. Lancet Psychiatry. 2025 Dec;12(12):906-920. doi: 10.1016/S2215-0366(25)00296-2. PMID 41233083
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, placebo-controlled, double-blind, multi-centre, multi-national, 26-week, parallel group trial, with a 4-week safety follow-up period. Participants had to complete the treatment and follow-up periods before they could enter the open label extension study.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the participants) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment sequence if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Iclepertin 10 mg | Placebo
Started | 306 | 305
Randomised to treatment | 306 | 305
Treated | 305 | 305
Completed | 267 | 267
Not Completed | 39 | 38
Not completed — Adverse Event | 14 | 15
Not completed — Burden of study procedures | 7 | 3
Not completed — Protocol deviation | 6 | 4
Not completed — Perceived lack of efficacy | 5 | 2
Not completed — Change of residence | 2 | 0
Not completed — Technical problems | 0 | 1
Not completed — Other than listed | 3 | 10
Not completed — No reason available | 1 | 3
Not completed — Patient randomised in error | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set (RS): included all patients who signed informed consent and were randomized into the trial, regardless of whether a patient was treated with trial medication. Patients randomized in error and discontinued from the study before the start of trial medication were excluded from the RS. Patients in the RS were analyzed under the randomized trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iclepertin 10 mg | Placebo | Total
Number analyzed (Participants) | 305 | 305 | 610
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.6 (8.5) | 35.5 (8.5) | 36.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 93 | 194
  Male | 204 | 212 | 416
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 89 | 78 | 167
  Not Hispanic or Latino | 199 | 213 | 412
  Unknown or Not Reported | 17 | 14 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 76 | 69 | 145
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 41 | 44 | 85
  White | 166 | 172 | 338
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Overall Composite T-score of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) After 26 Weeks of Treatment
Description: The change from baseline in MCCB (MATRICS Consensus Cognitive Battery) overall composite T-score at Week 26 is reported.
  This was analyzed using a mixed-effects model for repeated measurements (MMRM) comparing the change from baseline in MCCB overall composite T-score at Week 26 between iclepertin 10 mg daily and placebo. The MCCB comprises 10 tests to measure cognitive performance in 7 cognitive domains: speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The composite T-score is derived from the 7 cognitive domain T-scores. The T-score is standardized to the normative population with a mean of 50 and standard deviation of 10. A higher MCCB overall composite T-score indicates better cognition.
Time Frame: The MMRM model is a longitudinal analysis which incorporated values at screening, baseline and at Week 12 and Week 26. The data presented here represent the Least Squares Mean at Week 26.
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 305 | 305
T-score | 2.719 (0.3377) | 1.997 (0.3345)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; The model included fixed categorical effects of treatment at each visit and the stratification factor (screening MCCB overall composite T-score) and fixed effects for the continuous covariate of baseline at each visit. Visit was treated as a repeated measure with unstructured covariance structure for within-participant dependencies. The primary comparison was iclepertin 10 mg daily vs. placebo at Week 26; Test type: Superiority; p = 0.1291, Mixed Models Analysis; The Kenward-Roger method estimated denominator degrees of freedom and adjusted standard errors; Mean Difference (Net) = 0.722, 95% CI 2-sided [-0.211 to 1.656], Standard Error of Mean 0.4753 — Adjusted mean difference in overall composite T-score of the MCCB at Week 26 between the iclepertin 10 mg and the Placebo group

2. Secondary Outcome: Change From Baseline in SCoRS (Schizophrenia Cognition Rating Scale) Interviewer Total Score at Week 26
Description: SCoRS is a 20-item interview-based assessment of cognitive deficits and the degree to which they affect day-to-day functioning. Each item is rated on a 4-point scale, ranging from "No impairment" to "Severe Impairment", with higher ratings reflecting a greater degree of impairment. The SCoRS rater integrates information from separate patient and study partner interviews to generate a total score. SCoRS total score is between 20 and 80 where higher score values represent greater degree of impairment in day-to-day functions due to cognitive deficits. The total score was the sum of the 20 item scores. If six or more of the 20 items were missing, the total score was not derived and treated as missing for that participant at the visit, otherwise, missing items were imputed with the mean of the observed items for the purpose of total score calculation.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 305 | 305
Scores on a scale | -5.053 (0.4268) | -5.767 (0.4261)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; The model included the discrete fixed effects of treatment at each visit, fixed categorical covariate of the stratification factor using the screening MCCB overall composite T-score, and continuous fixed effects for the corresponding baseline endpoint value at each visit. Visit was treated as the repeated measure with an unstructured covariance structure to model the within-subject measurements. Subjects were considered as a random effect; Test type: Superiority; p = 0.2375, Mixed Models Analysis; The Kenward-Roger method estimated denominator degrees of freedom and adjusted standard errors; Mean Difference (Net) = 0.714, 95% CI 2-sided [-0.472 to 1.901], Standard Error of Mean 0.6042 — Adjusted mean difference in SCoRS at Week 26 between the iclepertin 10 mg and the Placebo group

3. Secondary Outcome: Change From Baseline in VRFCAT (Virtual Reality Functional Capacity Assessment Tool) Adjusted Total Time T-score at Week 26
Description: The VRFCAT is a virtual reality shopping trip performed on a tablet. The task has several linked and sequential scenarios, including matching a recipe to the content of kitchen cabinets, preparing a shopping list, taking the correct bus, shopping efficiently, and catching the correct return bus. These tasks are performed in a fixed sequence. The tool records the total amount of time taken to complete the sequence of tasks, adjusting for number of errors and forced progressions. A T-score is generated from this adjusted total time. The lower the adjusted total time T-score, the better is the patient's functional capacity. The T-score has a mean of 50 and a standard deviation of 10 in the normative population.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 305 | 305
T-score | 3.898 (0.7531) | 3.565 (0.7481)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7541, Mixed Models Analysis; The Kenward-Roger method estimated denominator degrees of freedom and adjusted standard errors; Mean Difference (Net) = 0.333, 95% CI 2-sided [-1.753 to 2.419], Standard Error of Mean 1.0620 — Adjusted mean difference in VRFCAT at Week 26 between the iclepertin 10 mg and the Placebo group

4. Secondary Outcome: Change From Screening Visit 1a to Week 24 in Patient Reported Experience of Cognitive Impairment in Schizophrenia (PRECIS) Total Score
Description: The Patient Reported Experience of Cognitive Impairment in Schizophrenia (PRECIS) score evaluates how cognitive difficulties impact the daily life of individuals with schizophrenia. It is composed of 28 items on a 5-category Likert scale (1=not at all/not at all hard, 5=very much/very hard), and the total score was derived by calculating the average score of the first 26 items, where higher scores indicate a worse patient experience. The questionnaire takes 5-15 minutes to complete and provides insights into cognitive impairment associated with schizophrenia (CIAS) impact.
Time Frame: The MMRM model is a longitudinal analysis which incorporated values at screening, and at Week 15 and Week 24. The data presented here represent the Least Squares Mean at Week 24.
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 305 | 305
Scores on a scale | -0.333 (0.0312) | -0.345 (0.031)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7769, Mixed Models Analysis; The Kenward-Roger method estimated denominator degrees of freedom and adjusted standard errors; Mean Difference (Net) = 0.012, 95% CI 2-sided [-0.074 to 0.099], Standard Error of Mean 0.0440 — Adjusted mean difference in PRECIS at Week 24 between the iclepertin 10 mg and the Placebo group

5. Secondary Outcome: Change From Baseline in the T-score of the Number of Correct Responses on Tower of London (ToL) at Week 26
Description: Change from baseline in the T-score of the number of correct responses on Tower of London at Week 26, using an analysis of covariance (ANCOVA) model, is reported. The Tower of London evaluates executive functions such as reasoning and problem-solving ability. It measures the number of correct responses in solving an exercise that involves moving colored balls to match a target configuration. The higher the ToL T-score, the better is the patient's cognitive function. A mean T-score of 50 and a standard deviation of 10 reflects the T-score in the normative population. The administration time was about 7 minutes.
Time Frame: Baseline and at Week 26
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Iclepertin 10 mg | Placebo
Number analyzed (Participants) | 305 | 305
T-Score | 0.148 (0.6446) | 1.283 (0.6433)
Statistical Analysis 1: Comparison: Iclepertin 10 mg vs Placebo; For change from baseline to Week 26 in the T-score of the number of correct responses on ToL, an analysis of covariance (ANCOVA) model including treatment, stratification factor of screening MCCB overall composite T-score (<30, ≥30), and baseline number of correct responses on ToL T-score were fitted to the data; Test type: Superiority; p = 0.2133, ANCOVA; Mean Difference (Net) = -1.135, 95% CI 2-sided [-2.925 to 0.654], Standard Error of Mean 0.9110 — Adjusted mean difference in ToL at Week 26 between the iclepertin 10 mg and the Placebo group

ADVERSE EVENTS:
Time Frame: Serious AEs and other AEs: From first dose of study drug to last dose over a 26-week treatment period, plus a 12-day residual effect period. All-cause mortality: From first drug administration till end of study over a 30-week observation period.
Description: The Treated Set (TS) included all patients who signed informed consent and were treated with at least one dose of the trial medication. Patients in the TS were analyzed under the actual trial medication received at randomization.
Arm/Group | Iclepertin 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/305 | 0/305
Serious Adverse Events (participants affected / at risk) | 11/305 | 16/305
Other Adverse Events (participants affected / at risk) | 73/305 | 59/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iclepertin 10 mg (N=305) | Placebo (N=305)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 1
Lymphadenitis bacterial (Infections and infestations) | 0 | 1
Pathogen resistance (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 2
Pneumocephalus (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 4 | 5
Suicidal ideation (Psychiatric disorders) | 0 | 4
Suicide attempt (Psychiatric disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iclepertin 10 mg (N=305) | Placebo (N=305)
Nasopharyngitis (Infections and infestations) | 22 | 17
Headache (Nervous system disorders) | 30 | 25
Somnolence (Nervous system disorders) | 18 | 15
Schizophrenia (Psychiatric disorders) | 20 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT04846881/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT04846881/SAP_001.pdf